CLINICAL TRIAL: NCT01510717
Title: Clinical Investigation of AcrySof® IQ ReSTOR® +2.5 D Multifocal Intraocular Lens (IOL) Model SN6AD2
Brief Title: Clinical Investigation of AcrySof® IQ ReSTOR® +2.5 D Multifocal Intraocular Lens (IOL) Model SN6AD2 [SV25T0]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-016
Record Dates: First submitted 2012-01-12; First posted 2012-01-16 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Cataracts
Keywords: Intraocular Lens; Monofocal; Multifocal
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal IOL (Experimental): AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0], bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]
- Monofocal IOL (Active Comparator): AcrySof® IQ Monofocal IOL Model SN60WF, bilateral implantation
  Interventions: Device: AcrySof® IQ Monofocal IOL Model SN60WF

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] — Multifocal IOL with extended secondary focal point implanted for long-term use over the lifetime of the cataract patient
  Arms: Multifocal IOL
Device: AcrySof® IQ Monofocal IOL Model SN60WF — Monofocal IOL implanted for long-term use over the lifetime of the cataract patient
  Arms: Monofocal IOL

SUMMARY:
The purpose of this study is to compare the safety and efficacy of an investigational multifocal intraocular lens (IOL) to an FDA-approved monofocal IOL.

DETAILED DESCRIPTION:
Participants 21 years and older in need of cataract extraction were consented and randomized in a 1:1 ratio at each investigative site to receive either the AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0] or the AcrySof® IQ Monofocal IOL Model SN60WF in both eyes. Each participant completed a preoperative examination of both eyes, implantation of IOL at the operative visit for each eye, and up to 7 postoperative visits, with monocular testing at Day 1-2, Day 7-14, and Day 30-60, and monocular and binocular testing at Day 120-180 following the second implantation. The first eye to be implanted was considered the primary eye. The second eye was implanted 7 and 30 days of the first. If the first eye was not implanted during surgery, the second eye was not eligible. If the second eye was not implanted during surgery, only the first eye was followed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral cataracts
* Willing and able to complete all required postoperative visits
* Calculated lens power within the available supply range
* Planned cataract removal by phacoemulsification
* Potential postoperative visual acuity of 0.2 logMAR or better in both eyes
* Preoperative astigmatism less than 1.0 diopter
* Clear intraocular media other than cataract in study eyes
* Preoperative Best Corrected Distance Visual Acuity (BCDVA) worse than 0.2 logMAR
* Able to undergo second eye surgery between 7 days and 30 days of the first eye surgery
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Previous refractive surgery
* Inflammation or edema of the cornea
* Optic nerve atrophy
* Pregnancy
* Current participation in another investigational drug or device study
* Other protocol-defined exclusion criteria may apply

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magda Michna, PhD, Study Director — Alcon Research

REFERENCES:
- [Derived] Williams JR, Kim HW, Crespi CM. Modeling observations with a detection limit using a truncated normal distribution with censoring. BMC Med Res Methodol. 2020 Jun 29;20(1):170. doi: 10.1186/s12874-020-01032-9. PMID 32600261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 15 investigative sites located in the United States.
Pre-assignment Details: Of the 409 participants enrolled, 80 were discontinued prior to randomization as screen failures and 9 were discontinued after randomization prior to implantation. This reporting group includes all participants with successful IOL implantation in at least 1 eye (320).
Groups:
- Multifocal IOL: AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]
- Monofocal IOL: AcrySof® IQ Monofocal IOL Model SN60WF
Period: Overall Study
Arm/Group | Multifocal IOL | Monofocal IOL
Started | 155 | 165
Completed | 153 | 160
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants with successful IOL implantation in at least 1 eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multifocal IOL | Monofocal IOL | Total
Number analyzed (Participants) | 155 | 165 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.64) | 69.4 (8.27) | 69.0 (8.95)
Age, Customized [Number; unit: participants]
  20-29 years | 1 | 0 | 1
  30-39 years | 2 | 0 | 2
  40-49 years | 2 | 3 | 5
  50-59 years | 18 | 12 | 30
  60-69 years | 53 | 62 | 115
  70-79 years | 65 | 71 | 136
  ≥80 years | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 97 | 193
  Male | 59 | 68 | 127
Region of Enrollment [Number; unit: participants]
  United States | 155 | 165 | 320

OUTCOME MEASURES:

1. Primary Outcome: Mean Photopic Monocular Distance Corrected VA (53 cm) at Day 120-180
Description: Visual acuity (VA) was tested monocularly (each eye separately) using the manifest refraction adjusted for optical infinity and the hand-held, 100% contrast, Early Treatment Diabetic Retinopathy Study (ETDRS) chart set at 53 centimeters (cm) on the nearpoint rod. VA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the primary eye.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in the primary eye.
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 155 | 165
Number analyzed (eyes) | 155 | 165
logMAR | 0.322 (0.014) | 0.512 (0.013)

2. Primary Outcome: Number of Cumulative and Persistent Adverse Events as Defined in IS EN ISO 11979-7:2006, up to Day 120-180
Description: Cumulative and persistent adverse events were collected. This outcome measure was prespecified for the multifocal IOL.
Time Frame: Day 0 first operative eye visit, up to Day 120-180 from second eye implantation
Population: This analysis population includes all participants with attempted IOL implantation in at least one eye (successful or aborted after contact with the eye).
Measure: Number; unit: adverse events
Units Other Than Participants: eyes
Arm/Group | Multifocal IOL
Number analyzed (Participants) | 155
Number analyzed (eyes) | 310
adverse events
  Cystoid macular oedema (cumulative) | 4
  Endophthalmitis (cumulative) | 0
  Hypopyon (cumulative) | 0
  Lens dislocated from posterior (cumulative) | 0
  Pupillary block (cumulative) | 0
  Retinal detachment (cumulative) | 0
  Secondary surgical intervention (cumulative) | 0
  Corneal stroma oedema (persistent) | 0
  Cystoid macular oedema (persistent | 2
  Iritis (persistent | 2
  Raised IOP requiring treatment (persistent) | 0

3. Primary Outcome: Photopic Contrast Sensitivity Without Glare at Day 120-180
Description: Contrast sensitivity (ie, the ability to detect objects by distinguishing them from their background) was assessed binocularly with the participant's best spectacle correction under photopic (bright) conditions at a distance of 8 feet at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd) using the Vector Vision CSV 1000 without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Scores of (-1) were set to missing; hence, the mean measures may be overestimated and the variability measures may be underestimated. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: The analysis population includes all participants with successful IOL implantation that had at least 1 postoperative visit, had no preoperative pathology or macular degeneration, and had no major protocol deviations at any time. Here n=number of participants with data for analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 133 | 137
logMAR
  3 cpd (n=131,133) | 1.676 (0.259) | 1.743 (0.203)
  6 cpd (n=130,133) | 1.816 (0.256) | 1.938 (0.251)
  12 cpd (n=129,132) | 1.460 (0.312) | 1.555 (0.312)
  18 cpd (n=130,131) | 0.970 (0.348) | 1.109 (0.325)

4. Secondary Outcome: Mean Photopic Monocular Best Corrected Distance VA (4 m) at Day 120-180
Description: VA was tested monocularly (each eye separately) using the correction obtained from the manifest refraction and 100% contrast, ETDRS charts at a distance of 4 meters. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the primary eye.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in the primary eye.
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 155 | 165
Number analyzed (eyes) | 155 | 165
logMAR | 0.025 (0.009) | 0.003 (0.009)

5. Secondary Outcome: Mean Photopic Monocular Distance Corrected Near VA at Standard Distance (40 cm) at Day 120-180
Description: VA was tested monocularly (each eye separately) using the manifest refraction adjusted for optical infinity and the hand-held, 100% contrast, ETDRS chart set at 40 cm on the nearpoint rod. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the primary eye.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in the primary eye.
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 155 | 165
Number analyzed (eyes) | 155 | 165
logMAR | 0.426 (0.014) | 0.632 (0.013)

6. Secondary Outcome: Overall Spectacle Independence Using SILVER Patient Reported Outcome (PRO) Questionnaire at Day 120-180
Description: Overall Spectacle Independence was rated using SILVER (Spectacle Independence Lens Vision Evaluation and Repurchase), a new patient reported outcome questionnaire. The participant was asked, "How often do you wear eyeglasses or contact lenses overall?"
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in at least 1 eye with data present.
Measure: Number; unit: participants
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 153 | 160
participants
  None of the time | 35 | 33
  Some of the time | 104 | 109
  Most of the time | 12 | 13
  All of the time | 2 | 5

7. Secondary Outcome: Near Spectacle Independence Using SILVER Patient Reported Outcome (PRO) Questionnaire at Day 120-180
Description: Near Spectacle Independence was rated using SILVER, a new patient reported outcome questionnaire. The participant was asked, "How often do you wear eyeglasses or contact lenses for seeing objects up close?"
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in at least 1 eye with data present.
Measure: Number; unit: participants
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 153 | 160
participants
  None of the time | 25 | 19
  Some of the time | 70 | 53
  Most of the time | 34 | 40
  All of the time | 24 | 48

8. Primary Outcome: Photopic Contrast Sensitivity With Glare at Day 120-180
Description: Contrast sensitivity was assessed binocularly with the participant's best spectacle correction under photopic (bright) conditions at a distance of 8 feet at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd) using the Vector Vision CSV 1000 with a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Scores of (-1) were set to missing; hence, the mean measures may be overestimated and the variability measures may be underestimated. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 133 | 137
logMAR
  3 cpd (n=130,131) | 1.608 (0.307) | 1.692 (0.274)
  6 cpd (n=117,125) | 1.684 (0.316) | 1.844 (0.309)
  12 cpd (n=117,127) | 1.334 (0.321) | 1.475 (0.336)
  18 cpd (n=119,128) | 0.914 (0.333) | 1.043 (0.361)

9. Primary Outcome: Mesopic Contrast Sensitivity Without Glare at Day 120-180
Description: Contrast sensitivity was assessed binocularly with the participant's best spectacle correction under mesopic (dim lighting) conditions at a distance of 8 feet at spatial frequencies of 1.5, 3, 6, and 12 cycles per degree (cpd) using the Vector Vision CSV 1000 without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Scores of (-1) were set to missing; hence, the mean measures may be overestimated and the variability measures may be underestimated. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 133 | 137
logMAR
  1.5 cpd (n=128,131) | 1.594 (0.224) | 1.622 (0.204)
  3 cpd (n=131,132) | 1.563 (0.267) | 1.618 (0.226)
  6 cpd (n=122,130) | 1.581 (0.296) | 1.673 (0.275)
  12 cpd (n=102,112) | 1.077 (0.363) | 1.208 (0.345)

10. Primary Outcome: Mesopic Contrast Sensitivity With Glare at Day 120-180
Description: Contrast sensitivity was assessed binocularly with the participant's best spectacle correction under mesopic conditions at a distance of 8 feet at spatial frequencies of 1.5, 3, 6, and 12 cpd using the Vector Vision CSV 1000 with a glare source. Raw scores from contrast sensitivity testing were transformed to log units. Scores of (-1) were set to missing; hence, the mean measures may be overestimated and the variability measures may be underestimated. A higher numeric value represents better contrast sensitivity.
Time Frame: Day 120-180 from second eye implantation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Multifocal IOL | Monofocal IOL
Number analyzed (Participants) | 133 | 137
logMAR
  1.5 cpd (n=127,129) | 1.536 (0.237) | 1.596 (0.238)
  3 cpd (n=128,130) | 1.542 (0.292) | 1.600 (0.296)
  6 cpd (n=114,126) | 1.543 (0.329) | 1.617 (0.277)
  12 cpd (n=90,105) | 1.043 (0.385) | 1.153 (0.375)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Feb 2012-Dec 2012).
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign, whether or not related to the investigational device. AEs were collected as solicited comments and as observations by the Investigator as outlined in the protocol. "At Risk" population for ocular AEs is included with unit of "eyes."
Groups:
- Pre-Treatment: All enrolled participants
- Multifocal IOL: All participants with attempted IOL implantation in at least one eye (successful or aborted after contact with the eye), AcrySof® IQ ReSTOR® +2.5 D Multifocal IOL Model SN6AD2 [SV25T0]
- Monofocal IOL: All participants with attempted IOL implantation in at least one eye (successful or aborted after contact with the eye), AcrySof® IQ Monofocal IOL Model SN60WF
Arm/Group | Pre-Treatment | Multifocal IOL | Monofocal IOL
Serious Adverse Events (participants affected / at risk) | 1/409 | 10/155 | 15/165
Other Adverse Events (participants affected / at risk) | 0/409 | 0/155 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pre-Treatment (N=409) | Multifocal IOL (N=155) | Monofocal IOL (N=165)
Cystoid macular oedema (First Implanted Eye) (Eye disorders) | 0 | 2 | 0
Intraocular pressure increased (First Implanted Eye) (Investigations) | 0 | 0 | 1
Open angle glaucoma (First Implanted Eye) (Eye disorders) | 0 | 0 | 1
Cataract operation complication (Second Implanted Eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1/163
Cystoid macular oedema (Second Implanted Eye) (Eye disorders) | 0 | 2 | 0/163
Device dislocation (Second Implanted Eye) (General disorders) | 0 | 0 | 1/163
Eye operation (Second Implanted Eye) (Surgical and medical procedures) | 0 | 0 | 1/163
Intraocular injection (Second Implanted Eye) (Surgical and medical procedures) | 0 | 0 | 1/163
Intraocular pressure increased (Second Implanted Eye) (Investigations) | 0 | 0 | 1/163
Iritis (Second Implanted Eye) (Eye disorders) | 0 | 0 | 1/163
Open angle glaucoma (Second Implanted Eye) (Eye disorders) | 0 | 0 | 1/163
Retinal vein occlusion (Second Implanted Eye) (Eye disorders) | 0 | 0 | 1/163
Surgical procedure repeated (Second Implanted Eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1/163
Wound complication (Second Implanted Eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1/163
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1 | 0
Incisional hernia gangrenous (Infections and infestations) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.